CLINICAL TRIAL: NCT02157194
Title: Endobronchial Ultrasound-transbronchial Needle Aspiration (EBUS-TBNA) Sample Division
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Kaid Darwiche, Senior Physician Interventional Pneumology, University Hospital, Essen
Other Study IDs: RLK-EBUS-2; 11-4921-BO (Other: EC UK Essen)
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
EBUS-TBNA specimen are used for lung cancer diagnosing and staging, as well for molecular analysis. The purpose of this study is to evaluate if samples from on lymph node site can be divided for diagnosis and molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lung cancer
* enlarged mediastinal or hilar lymph nodes (>10 mm)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suspected to have lung cancer and enlarged mediastinal lymph nodes
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of lung cancer diagnosis | 6 month
  We aim to evaluate if splitting the obtained specimen will have an impact on lung cancer diagnosis performed by histopathologic analysis

SECONDARY OUTCOMES:
Percentage of successful performed molecular RNA based analysis | 3 month
  We will analyse the second half of the sample regarding molecular analysis. RNA concentration and RNA integrity score will be assessed before a new RNA based test will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruhrlandklinik-UK Essen, Essen, Germany